CLINICAL TRIAL: NCT01752699
Title: Methadone in Post-Herpetic Neuralgia Pain
Acronym: NPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPH
Record Dates: First submitted 2012-12-11; First posted 2012-12-19 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Post-herpetic Neuralgia
Keywords: neuropathic pain,; post-herpetic neuralgia,; methadone,
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methadone (Experimental): in this arm patients will take methadone 5mg.
  Interventions: Drug: Methadone
- Placebo (Experimental): in this arm patients will take placebo pills.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methadone — patients with post-herpetic neuralgia take methadone or placebo to treat pain symptoms.
  Arms: Methadone
Drug: Placebo — patients with post-herpetic neuralgia take placebo to treat the pain symptoms.
  Arms: Placebo

SUMMARY:
Neuropathic pain is a common condition and affecting 40 to 70% of the general population. Post-herpetic neuralgia is a condition almost complex and requires a multi modal treatment. Aim: This is a pilot proof-of-principle study designed to evaluate the use of low-dose methadone in post-herpetic neuralgia patients who remained refractory after first and second line treatment for post-herpetic neuralgia (PHN) and had indication for the association of an opioid agent to their current drug regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic (>6 months) symptomatic PHN
* with visual analogical scale >40/100mm
* use of first and second line drugs (tricyclic antidepressants, venlafaxine and gabapentinoids)

Exclusion Criteria:

* Don't full the criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1998-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline Pain | baseline (visit inclusion) and three moths latter
  Assessing by verbal analog scale (VAS)

REFERENCES:
- [Derived] Teixeira MJ, Okada M, Moscoso AS, Puerta MY, Yeng LT, Galhardoni R, Tengan S, Andrade DC. Methadone in post-herpetic neuralgia: A pilot proof-of-concept study. Clinics (Sao Paulo). 2013 Jul;68(7):1057-60. doi: 10.6061/clinics/2013(07)25. PMID 23917673